CLINICAL TRIAL: NCT05600452
Title: Comparison of a Novel Condensed Heat Acclimation Programme With a Traditional Longer-term Heat Acclimation Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: Coventry University (Other); Teesside University (Other)
Responsible Party: Principal Investigator, Jo Corbett, Reader in Environmental Physiology, University of Portsmouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1017/MoDREC/19
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Heat Stress
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Parallel groups design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional heat acclimation (Active Comparator): The traditional heat acclimation programme will consist of daily 75-minute heat exposures for eight consecutive days
  Interventions: Other: Heat acclimation
- Condensed heat acclimation (Experimental): The condensed heat acclimation programme will consist of two consecutive days with four, 75-minute heat exposures undertaken on each day
  Interventions: Other: Heat acclimation

INTERVENTIONS:
Other: Heat acclimation — Repeated heat exposures with light exercise sufficient to elevate deep body temperature to ~ 38.5C

SUMMARY:
Repeated exposure to heat in a laboratory setting (acclimation) elicits a range of adaptations, which reduce heat illness risk and increase work capacity in the heat. Traditional approaches to heat acclimation require daily heat exposures of 1 to 2 hours over ~7 to 10 consecutive days. Heat acclimation approaches which reduce the number of days to achieve acclimation may have utility. The primary purpose of the proposed research is to determine whether it is possible to achieve a similar degree of heat acclimation to that seen with a traditional longer-term heat acclimation approach by increasing the frequency of heat exposure, utilising multiple daily heat exposures over a smaller number of days. Secondary aims of the research are to examine whether heat acclimation provides cross-adaptation to a hypoxic stressor and whether heat acclimation improves aerobic fitness.

DETAILED DESCRIPTION:
Individuals are often required to operate in adverse conditions and may be exposed to prolonged periods of high ambient heat and humidity. High environmental temperatures impair work capacity and increase heat-illness risk. Repeated exposure to heat in a laboratory setting (acclimation) elicits a range of adaptations, which reduce heat illness risk and increase work capacity in the heat. However, traditional approaches to heat acclimation are time consuming, typically requiring daily heat exposures of 1 to 2 hours over ~7 to 10 consecutive days. This can be logistically difficult to implement and impractical, particularly in situations where an individual must be rapidly deployed. Therefore, heat acclimation approaches which reduce the number of days to achieve acclimation may have utility. In addition, recent research studies have suggested that adaptation to heat may improve tolerance to hypoxia (cross-adaptation) and improve aerobic fitness; these effects may also be beneficial in a military context. Therefore, the primary purpose of the proposed research is to determine whether it is possible to achieve a similar degree of heat acclimation to that seen with a traditional longer-term heat acclimation approach by increasing the frequency of heat exposure, utilising multiple daily heat exposures over a smaller number of days. Secondary aims of the research are to examine whether heat acclimation provides cross-adaptation to a hypoxic stressor and whether heat acclimation improves aerobic fitness. Heat acclimation will be evaluated using a range of whole-body (cardiovascular, thermoregulatory, psychophysiological) and biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Physically active and healthy as determined by pre-participation health screening questionnaire.
* Free of COVID-19 symptoms (loss or change in sense of smell or taste, fever and new, continuous cough) as determined by pre-screening questionnaire.
* Resting diastolic blood pressure between 60 and 90 mmHg; resting systolic blood pressure between 90 and 150 mmHg A resting ECG is required if: individuals are over 30 years of age; they are unfamiliar with exercise of a maximal nature; they have a family history of adverse cardiac events. The ECG is to be reviewed by the Independent Medical Officer.

Exclusion Criteria:

* Current smokers
* Recent (< 3 months) participation in a formal heat acclimation regimen, or regular frequent heat exposures that may render the participant partially heat acclimated (other than regular exercise)
* Recent (< 3 months) high altitude (>1 500m ) sojourn that may render the participant partially altitude acclimated
* Diagnosed cardiovascular, metabolic or respiratory conditions (excluding asthma)
* Prior history of heat illness
* Prior history of collapse or intolerance with exposure to altitude
* Recent blood donation (within 3 months of commencing study)
* Baseline serum sodium level <135 mmol.L-1
* Any other extant medical condition which may be exacerbated by participation
* Participants with inadequate understanding of English.
* Any volunteers who are currently participating in any other research studies which may influence their responses or the results obtained

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Reduction in the peak deep body temperature | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Rectal temperature measurement during a heat stress test

SECONDARY OUTCOMES:
Reduction in the resting deep body temperature | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Rectal temperature measurement during a heat stress test
Reduction in the peak mean body temperature | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Weighted rectal and mean skin temperature measurement during a heat stress test
Reduction in the resting mean body temperature | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Weighted rectal and mean skin temperature measurement during a heat stress test
Increased plasma volume | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Change in plasma volume calculated from resting haemoglobin and haematocrit prior to a heat stress test
Increased sweating rate | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Sweating rate calculated from change in nude body mass and accounting for fluid consumption during a heat stress test
Reduced sweat sodium concentration | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Sweating sodium concentration assessed from sweat collected in a custom sweat patch on the back during a heat stress test
Reduced exercise heart rate | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Heart rate measured using chest telemetry during a heat stress test
Increased resting intracellular heat shock protein 70 content | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Assessed in peripheral blood mononuclear cells obtained before a heat stress test
Increased post heat stress intracellular heat shock protein 70 content | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Assessed in peripheral blood mononuclear cells obtained after a heat stress test
Increased resting intracellular heat shock protein 90 alpha content | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Assessed in peripheral blood mononuclear cells obtained before a heat stress tests
Increased post heat stress intracellular heat shock protein 90 alpha content | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Assessed in peripheral blood mononuclear cells obtained after a heat stress tests
Maximal oxygen uptake | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Highest rate of oxygen uptake during graded cycling exercise
Lactate threshold | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Power output at 4 mmol.L-1 blood lactate during graded cycling exercise
Gross mechanical efficiency | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Percentage ratio of external work achieved compared to the total energy expenditure during graded cycling exercise below the lactate threshold
Peak power output | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Highest power output achieved during exhaustive cycling exercise
Peripheral oxygen saturation during exposure to hypoxia | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Assessed using ear or finger tip pulse oximetry during a hypoxic tolerance test
Heart rate during exposure to hypoxia | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Assessed using chest telemetry during a hypoxic tolerance test
Minute ventilation during exposure to hypoxia | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Expire volume of air per minute during a hypoxic tolerance test
Plasma neutrophil gelatinase-associated lipocalin | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Concentration change pre to post heat stress test
Urine neutrophil gelatinase-associated lipocalin | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Concentration change pre to post heat stress test
Plasma kidney injury molecule-1 | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Concentration change pre to post heat stress test
Urine kidney injury molecule-1 | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Concentration change pre to post heat stress test
Tissue inhibitor of metalloproteinase 2 | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Urine concentration change pre to post heat stress test
Insulin-like growth factor-binding protein 7 | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Urine concentration change pre to post heat stress test
Intestinal fatty acid binding protein | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Serum concentration change pre to post heat stress test
Soluble cluster of differentiation 14 | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Plasma concentration change pre to post heat stress test
Lipopolysaccharide binding protein | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Plasma concentration change pre to post heat stress test
Interleukin-6 | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Plasma concentration change pre to post heat stress test
Cortisol | Pre heat acclimation intervention (up to 1 week) to post heat acclimation intervention (up to 1 week)
  Plasma concentration change pre to post heat stress test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be published as measures of central tendency and dispersion (e.g. Mean and Standard deviation)